CLINICAL TRIAL: NCT02903823
Title: Intrathecal (IT) Baclofen Drug Distribution Pilot Study
Brief Title: Intrathecal (IT) Baclofen Drug Distribution
Acronym: ITB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Peter Konrad, MD, PhD, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 151399
Record Dates: First submitted 2016-08-26; First posted 2016-09-16 (Estimated); Results first posted 2021-04-27 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Muscle Spasticity
Keywords: spinal cord injury; cerebral palsy; stroke
MeSH Terms: conditions — Muscle Spasticity; Spinal Cord Injuries; Cerebral Palsy; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Baclofen injection at designated spinal level (Experimental): Days 2,3,4,5 a baclofen injection bolus will be given in the catheter, located at C4, T4, T10 and L2 respectively. Effect of baclofen injection (50 microgram bolus) upon rigidity will be assessed manually using the Modified Ashworth rating score for selected upper and lower extremities.
  Interventions: Drug: Baclofen bolus injection

INTERVENTIONS:
Drug: Baclofen bolus injection — A baclofen bolus injection (50 micrograms) will be administered daily after the patient returns from radiology to position catheter injection location. The injection may be given at C4, T4, T10 or L2 spinal locations depending on the catheter tip location.
  Other Names: Injection of baclofen bolus

SUMMARY:
The goal of this pilot study to determine whether there is a significant therapeutic advantage to place the ITB catheter within the cervical, thoracic or lumbar region of the spine. It is also a goal of this pilot study to determine whether the origin of spasticity influences the effect of Lioresal Intrathecal (baclofen injection) on ITB catheters located in the cervical, thoracic or lumbar regions of the spine. The investigators propose to study the impact of catheter location on the reduction in spasticity within a group of patients who are scheduled for ITB trial.

DETAILED DESCRIPTION:
While ITB therapy is commonly recommended for treatment of severe spasticity due to a variety of diseases, the location of optimal drug (baclofen) delivery has not been defined in a controlled study. Furthermore, the cost of pharmacological management in these patients is significant, and optimal location for drug delivery through an implantable drug pump may have significant impact on the cost burden of maintenance refills. It is the goal of this pilot study to determine whether there is a significant therapeutic advantage to place the ITB catheter within the cervical, thoracic or lumbar region of the spine. It is also a goal of this pilot study to determine whether the origin of spasticity influences the effect of Lioresal Intrathecal (baclofen injection) on ITB catheters located in the cervical, thoracic or lumbar regions of the spine. The investigators propose to study the impact of catheter location on the reduction in spasticity within a group of patients who are scheduled for ITB trial. In studying the impact of catheter location among patients with spinal versus cerebral origin of spasticity, the disease origin may also have a significant impact on baclofen dosing relative to the placement of the catheter.

In addition, the pharmacokinetic half-life and the variability of intrathecal baclofen is poorly understood as data is limited. In order to provide initial data regarding CSF baclofen washout, samples of spinal fluid obtained just prior to- and following IT baclofen administration will be obtained for delayed analysis. The results of these pharmacological analysis may refine the understanding of how quickly baclofen is distributed from a given catheter location, and whether it is affected by catheter location or disease origin. Since multiple catheter locations will be studied within a given patient, it also affords the opportunity to sample small amounts of CSF at key anatomical sites along the spinal axis as a secondary objective.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with spasticity from spinal origin (spinal cord injury)
2. Adult patients with spasticity of cerebral origin (cerebral palsy and cerebrovascular accident)
3. Adult women of child bearing age with a negative pregnancy test

Exclusion Criteria:

1. Patients with spasticity from Multiple sclerosis
2. Pregnant women
3. Patients under the age of 18 years
4. Patients over the age of 50
5. Patients who are unable to have an MRI scan of the total spine
6. Patients with spinal deformity that would prevent easy access to the lumbar intrathecal space
7. Patients who have an allergic reaction to IT baclofen
8. Patients who have significant headache from CSF withdrawal
9. Patients who have intradural blockage that prevents advancing the IT catheter to the level of C4

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-04-22 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Penn RD. Catheter implant systems for intrathecal drug delivery. J Neurosurg. 1996 Apr;84(4):713. doi: 10.3171/jns.1996.84.4.0713a. No abstract available. PMID 8613874
- [Background] Kroin JS, Ali A, York M, Penn RD. The distribution of medication along the spinal canal after chronic intrathecal administration. Neurosurgery. 1993 Aug;33(2):226-30; discussion 230. PMID 7690122
- [Background] Grabb PA, Guin-Renfroe S, Meythaler JM. Midthoracic catheter tip placement for intrathecal baclofen administration in children with quadriparetic spasticity. Neurosurgery. 1999 Oct;45(4):833-6; discussion 836-7. doi: 10.1097/00006123-199910000-00020. PMID 10515478
- [Background] Albright AL. Technique for insertion of intraventricular baclofen catheters. J Neurosurg Pediatr. 2011 Oct;8(4):394-5. doi: 10.3171/2011.7.PEDS11211. PMID 21961547
- [Background] Coffey JR, Cahill D, Steers W, Park TS, Ordia J, Meythaler J, Herman R, Shetter AG, Levy R, Gill B, et al. Intrathecal baclofen for intractable spasticity of spinal origin: results of a long-term multicenter study. J Neurosurg. 1993 Feb;78(2):226-32. doi: 10.3171/jns.1993.78.2.0226. PMID 8421205
- [Background] Albright AL, Turner M, Pattisapu JV. Best-practice surgical techniques for intrathecal baclofen therapy. J Neurosurg. 2006 Apr;104(4 Suppl):233-9. doi: 10.3171/ped.2006.104.4.233. PMID 16619633

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects recruited through Vanderbilt University Adult Neurosurgery group in Nashville, TN.
  Intent was to enroll subjects until 20 completed the study. Hence 7 more subjects were enrolled than completed. That makes 27 that started the study and 20 completed it.
  .
Period: Overall Study
Arm/Group | Baclofen Injection at Designated Spinal Level
Started | 27 (First subject enrollment)
Completed | 20
Not Completed | 7
Not completed — Physician Decision | 5
Not completed — Could not advance catheter | 1
Not completed — Catheter dislodgement | 1

BASELINE CHARACTERISTICS:
Population: Subjects who were assessed after initial catheter placement with baseline MAS and spasm scores.
Arm/Group | Baclofen Injection at Designated Spinal Level
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 43 [20 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Subjects Experiencing Maximal MAS Change From Baseline - Spasticity of Cerebral Origin
Description: The Modified Ashworth Scale (MAS) is a 6-point scale (Standard MAS scale values: "0, 1, 1.5, 2, 3, or 4") used to evaluate spasticity based on grading muscle tone by moving joints. The MAS scores in this cohort are measured in biceps, triceps and forearm flexor muscles in upper extremities; and quadriceps, hamstrings and gastrocnemius muscles in lower extremities. The score ranges from 0 (no increase in muscle tone) to 4 (affected part(s) rigid in flexion or extension). Improvement in spasticity was a reduction in MAS score by 1 point across a joint tested. Maximal MAS change is the sum of MAS score reduction in all four limbs tested.
  This outcome looks at subjects with spasticity of cerebral origin.
Time Frame: Baseline to 6 hours post-injection
Population: Subjects with pre-surgical diagnosis of spasticity of cerebral origin.
Measure: Count of Participants; unit: Participants
Groups:
- Subjects With Max MAS Change: Days 2,3,4,5 a baclofen injection bolus will be given in the catheter, located at C4, T3, T10 and L2 respectively. Effect of baclofen injection (50 microgram bolus) upon rigidity will be assessed manually using the Modified Ashworth rating score for selected upper and lower extremities.
  Baclofen bolus injection: A baclofen bolus injection (50 micrograms) will be administered daily after the patient returns from radiology to position catheter injection location. The injection may be given at C4, T4, T10 or L2 spinal locations depending on the catheter tip location.
Arm/Group | Subjects With Max MAS Change
Number analyzed (Participants) | 20
Participants
  Cervical level 4 injection site | 8
  Thoracic level 3 injection site | 7
  Thoracic level 10 injection site | 3
  Lumbar lever 2 injection site | 3

2. Primary Outcome: Subjects Experiencing Maximal MAS Change From Baseline - Spasticity of Spinal Origin
Description: The Modified Ashworth Scale (MAS) is a 6-point scale (Standard MAS scale values: "0, 1, 1.5, 2, 3, or 4") used to evaluate spasticity based on grading muscle tone by moving joints. The MAS scores in this cohort are measured in biceps, triceps and forearm flexor muscles in upper extremities; and quadriceps, hamstrings and gastrocnemius muscles in lower extremities. The score ranges from 0 (no increase in muscle tone) to 4 (affected part(s) rigid in flexion or extension). Improvement in spasticity was a reduction in MAS score by 1 point across a joint tested. Maximal MAS change is the sum of MAS score reduction in all four limbs tested.
  This outcome looks at subjects with spasticity of spinal origin.
Time Frame: Baseline to 6 hours post-injection
Measure: Count of Participants; unit: Participants
Groups:
- Subjects With MAS Change - Based on Site of Injection: Days 2,3,4,5 a baclofen injection bolus will be given in the catheter, located at C4, T3, T10 and L2 respectively. Effect of baclofen injection (50 microgram bolus) upon rigidity will be assessed manually using the Modified Ashworth rating score for selected upper and lower extremities.
  Baclofen bolus injection: A baclofen bolus injection (50 micrograms) will be administered daily after the patient returns from radiology to position catheter injection location. The injection may be given at C4, T4, T10 or L2 spinal locations depending on the catheter tip location.
Arm/Group | Subjects With MAS Change - Based on Site of Injection
Number analyzed (Participants) | 20
Participants
  Cervical spine level 4 injection site | 4
  Thoracic level 3 injection site | 2
  Thoracic level 10 injection site | 5
  Lumbar level 2 injection site | 3

ADVERSE EVENTS:
Time Frame: 5 days
Groups:
- Baclofen Injection at Designated Spinal Level: Days 2,3,4,5 a baclofen injection bolus will be given in the catheter, located at C4, T3, T10 and L2 respectively. Effect of baclofen injection (50 microgram bolus) upon rigidity will be assessed manually using the Modified Ashworth rating score for selected upper and lower extremities.
  Baclofen bolus injection: A baclofen bolus injection (50 micrograms) will be administered daily after the patient returns from radiology to position catheter injection location. The injection may be given at C4, T4, T10 or L2 spinal locations depending on the catheter tip location.
Arm/Group | Baclofen Injection at Designated Spinal Level
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 1/27
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baclofen Injection at Designated Spinal Level (N=27)
Catheter dislodgement (Nervous system disorders) | 1 (1) — catheter dislodged from location during manipulation in middle of study

LIMITATIONS AND CAVEATS:
Small number of subjects. Non-randomized trial. Inter-rater variability of assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT02903823/Prot_SAP_000.pdf